CLINICAL TRIAL: NCT04698941
Title: Clinical Study of Albumin Paclitaxel With or Without Simvastatin in Treating Extensive-Stage Small Cell Lung Cancer Patients Relapsed From First-line Chemotherapy
Brief Title: Combined Simvastatin and Albumin Paclitaxel in Treating ES-SCLC Patients Relapsed From 1st Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Yayi He, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020LY021
Record Dates: First submitted 2020-12-30; First posted 2021-01-07 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Small Cell Lung Cancer
Keywords: ES-SCLC; Chemo-resistance; Simvastatin
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Simvastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simvastatin + Albumin Paclitaxel (Experimental): received intravenous infusions of Paclitaxel 260 milligrams per square meter (mg/m^2) on Day 1 of every 21-day cycle (4 cycles) in combination with oral simvastatin (20mg daily) (10 months)
  Interventions: Drug: Albumin Paclitaxel; Drug: Simvastatin
- Albumin Paclitaxel (Active Comparator): received intravenous infusions of Paclitaxel 260 milligrams per square meter (mg/m^2) on Day 1 of every 21-day cycle (4 cycles)
  Interventions: Drug: Albumin Paclitaxel

INTERVENTIONS:
Drug: Albumin Paclitaxel — Albumin Paclitaxel intravenous infusion was administered at a dose of 260 mg/m^2 on Day 1 of each 21-day cycle.
Drug: Simvastatin — 20mg daily oral tablet taken.
  Other Names: Simvastatin Tablets
  Arms: Simvastatin + Albumin Paclitaxel

SUMMARY:
This Phase II study was designed to evaluate the safety and efficacy of albumin paclitaxel in combination with simvastatin compared with treatment with albumin paclitaxel alone in ES-SCLC patients relapsed from first-line chemotherapy. Participants will be divided in a 1:1 ratio to receive either albumin paclitaxel (4 cycles) + simvastatin (10 months) or albumin paclitaxel (4 cycles) until progressive disease (PD) as assessed by the investigator using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) or symptomatic deterioration.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I.To assess disease control rate (DCR) after treatment.

SECONDARY OBJECTIVES:

I.To assess best overall response rate (ORR) after treatment. II.To evaluate the progression-free survival (PFS) of patients with extensive stage-small cell lung cancer (ES-SCLC) treated with albumin paclitaxel + simvastatin or with albumin paclitaxel alone.

III.To estimate overall survival (OS) of patients with ES-SCLC. IV. To evaluate the toxicity profile of albumin paclitaxel + simvastatin.

EXPLORATORY OBJECTIVES:

I.To evaluate biomarkers correlatives. II.To explore the mechanism of albumin paclitaxel + simvastatin in the treatment of chemotherapy-resistant participants with ES-SCLC.

OUTLINE: Patients are divided into two arms. ARM A: Participants received intravenous infusions of albumin paclitaxel 260 milligrams per square meter (mg/m^2) on Day 1 of every 21-day cycle in combination with oral simvastatin (20mg daily) until persistent radiographic PD as assessed by the investigator using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) or symptomatic deterioration.

ARM B:Participants received intravenous infusions of albumin paclitaxel 260 mg/m^2 alone on Day 1 of every 21-day cycle until persistent radiographic PD, symptomatic deterioration, intolerable toxicity, withdrawal of consent, death, or study termination by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be volunteered to participate in the clinical trial. Patients must sign the informed Consent form (ICF) and be willing to follow and be able to complete all test procedures.
2. Histologically or cytologically confirmed ES-SCLC (per the Veterans Administration Lung Study Group [VALG] staging system).
3. No patients with resectable or radical radiotherapy lung cancer.
4. Patient must have no Epidermal Growth Factor Receptor (EGFR) mutation, Anaplastic lymphoma kinase (ALK) rearrangement, or ROS proto-oncogene 1 , receptor tyrosine kinase(ROS1) rearrangement.
5. Patient must be at least resistant to the first-line chemotherapy.
6. Patients must have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
7. Patients can tolerate chemotherapy.

Exclusion Criteria:

1. Unclear diagnosis of SCLC.
2. Resectable or radical radiotherapy SCLC.
3. Contraindicated chemotherapy.
4. Undergoing other active malignancies within 5 years or at the same time.Patients with localized curable tumors, such as basal cell carcinoma, squamous cell carcinoma, superficial bladder carcinoma, prostate carcinoma in situ, cervical carcinoma in situ, or breast carcinoma in situ, will not be excluded.
5. Positive test result for human immunodeficiency virus (HIV).
6. Positive test result for active tuberculosis.
7. Live vaccine was administered within 28 days of initial administration. Inactivated viral vaccines for seasonal influenza are allowed, except for live attenuated intranasal vaccines.
8. Pregnant or lactating women.
9. A history of psychotropic substance abuse, drug abuse, or alcoholism.
10. Other factors assessed by the sponsors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-25 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) | 6 weeks
  To assess disease control rate (DCR) after treatment.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 6 weeks
  To assess best overall response rate (ORR) after treatment.
Progression-free survival (PFS) | 12 weeks
  To evaluate the progression-free survival (PFS) of patients with extensive stage small cell lung cancer (ES-SCLC) treated with paclitaxel + simvastatin or with paclitaxel alone.
Overall survival (OS) | 24 weeks
  To estimate overall survival (OS) of patients with ES-SCLC.
Number of participants with treatment-related adverse events (AE) as assessed by CTCAE v4.0 | 24 weeks
  To evaluate the toxicity profile.

CONTACTS AND LOCATIONS:
Overall Officials: Yayi He, Doctor, Principal Investigator — Shanghai Pulmonary Hospital, Tongji University
Locations (2):
- China (2):
  - CAS Center for Excellence in Molecular Cell Science, Shanghai Institute of Biochemistry and Cell Biology, Chinese Academy of Sciences, Shanghai, Shanghai Municipality
  - Shanghai pulmonary hospital, Tongji University, Shanghai, Shanghai Municipality

REFERENCES:
- [Background] Goldman JW, Dvorkin M, Chen Y, Reinmuth N, Hotta K, Trukhin D, Statsenko G, Hochmair MJ, Ozguroglu M, Ji JH, Garassino MC, Voitko O, Poltoratskiy A, Ponce S, Verderame F, Havel L, Bondarenko I, Kazarnowicz A, Losonczy G, Conev NV, Armstrong J, Byrne N, Thiyagarajah P, Jiang H, Paz-Ares L; CASPIAN investigators. Durvalumab, with or without tremelimumab, plus platinum-etoposide versus platinum-etoposide alone in first-line treatment of extensive-stage small-cell lung cancer (CASPIAN): updated results from a randomised, controlled, open-label, phase 3 trial. Lancet Oncol. 2021 Jan;22(1):51-65. doi: 10.1016/S1470-2045(20)30539-8. Epub 2020 Dec 4. PMID 33285097
- [Background] Gelsomino F, Tiseo M, Barbieri F, Riccardi F, Cavanna L, Frassoldati A, Delmonte A, Longo L, Dazzi C, Cinieri S, Colantonio I, Sperandi F, Lamberti G, Brocchi S, Tofani L, Boni L, Ardizzoni A. Phase 2 study of NAB-paclitaxel in SensiTivE and refractory relapsed small cell lung cancer (SCLC) (NABSTER TRIAL). Br J Cancer. 2020 Jul;123(1):26-32. doi: 10.1038/s41416-020-0845-3. Epub 2020 Apr 29. PMID 32346071
- [Background] Chen Y, Li X, Zhang R, Xia Y, Shao Z, Mei Z. Effects of statin exposure and lung cancer survival: A meta-analysis of observational studies. Pharmacol Res. 2019 Mar;141:357-365. doi: 10.1016/j.phrs.2019.01.016. Epub 2019 Jan 11. PMID 30641276
- [Background] Khanzada UK, Pardo OE, Meier C, Downward J, Seckl MJ, Arcaro A. Potent inhibition of small-cell lung cancer cell growth by simvastatin reveals selective functions of Ras isoforms in growth factor signalling. Oncogene. 2006 Feb 9;25(6):877-87. doi: 10.1038/sj.onc.1209117. PMID 16170339
- [Background] Holstein SA, Hohl RJ. Synergistic interaction of lovastatin and paclitaxel in human cancer cells. Mol Cancer Ther. 2001 Dec;1(2):141-9. PMID 12467231